CLINICAL TRIAL: NCT02040428
Title: A Single-blinded, Randomized, Controlled, Comparative Phase III Study Evaluating the Safety and Effectiveness of EVARREST™ Fibrin Sealant Patch as an Adjunct to Hemostasis During Cardiovascular Surgery
Brief Title: The Fibrin Pad CV Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS-13-004; 2013-003464-31 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Diseases; Fibrin Sealant; Hemostatics; Coagulants
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EVARREST™ Fibrin Sealant Patch (Experimental): EVARREST™ Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Interventions: Biological: EVARREST™ Fibrin Sealant Patch
- Topical hemostat (Active Comparator): Equine collagen with Human Fibrinogen and Human Thrombin
  Interventions: Biological: Topical hemostat

INTERVENTIONS:
Biological: EVARREST™ Fibrin Sealant Patch
  Arms: EVARREST™ Fibrin Sealant Patch
Biological: Topical hemostat
  Arms: Topical hemostat

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the EVARREST™ Fibrin Sealant Patch as an adjunct to hemostasis during cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age, requiring an elective or urgent, open aortic surgical procedure utilizing cardiopulmonary bypass. Subjects in Japan between ≥18 and <20 years of age will require consent by the subject's legal representative
* Subjects must be willing to participate in the study and provide written informed consent.
* Presence of an appropriate Target Bleeding Site (TBS) along the anastomotic suture line, involving a synthetic aortic graft, as identified intra-operatively by the investigator;

Exclusion Criteria:

* Subjects with known intolerance to blood products or to one of the components of the study product or unwilling to receive blood products;
* Exposure to another investigational drug or device in a clinical trial within 30 days prior to surgery or anticipated in the 60 day follow up period after surgery.
* Female subjects who are pregnant or nursing.
* TBS is from a large defects in visible arteries or veins where the injured vascular wall requires repair and maintenance of vessel patency or where there would be persistent exposure of EVARREST™ Fibrin Sealant Patch to blood flow and/or pressure during absorption of the product;
* TBS with major arterial bleeding requiring suture or mechanical ligation;
* TBS involves an expanded polytetrafluoroethylene (ePTFE) graft
* TBS within an actively infected field;
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine;
* Subjects with any intra-operative findings identified by the investigator that may preclude conduct of the study procedure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (24):
- United States (9):
  - Clinical Investigation Site #15, Atlanta, Georgia
  - Clinical Investigation Site #14, Indianapolis, Indiana
  - Clinical Investigation Site #16, Baltimore, Maryland
  - Clinical Investigation Site #21, Bethesda, Maryland
  - Clinical Investigation Site #17, St Louis, Missouri
  - Clinical Investigation Site #10, Paterson, New Jersey
  - Clinical Investigation Site #12, New York, New York
  - Clinical Investigation Site #20, Philadelphia, Pennsylvania
  - Clinical Investigation Site #18, Houston, Texas
- Australia (5):
  - Clinical Investigation Site #72, Camperdown, New South Wales
  - Clinical Investigation Site #73, Sydney, New South Wales
  - Clinical Investigation Site #71, Brisbane, Queensland
  - Clinical Investigation Site #74, Bedford Park, South Australia
  - Clinical Investigation Site #70, Melbourne, Victoria
- Clinical Investigation Site #40, Ghent, Belgium
- Japan (3):
  - Clinical Investigation Site #82, Kanagawa, Isehara-shi
  - Clinical Investigation Site #81, Saitama, Saitama-shi
  - Clinical Investigation Site #80, Osaka, Suita-shi
- United Kingdom (6):
  - Clinical Investigation Site #33, Bristol, England
  - Clinical Investigation Site #35, Cottingham, England
  - Clinical Investigation Site #34, Manchester, England
  - Clinical Investigation Site #32, Aberdeen, Scotland
  - Clinical Investigation Site #31, Clydebank, Scotland
  - Clinical Investigation Site #30, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from January 13, 2014 through September 23, 2015 at hospitals and medical centers throughout the United States, United Kingdom, Belgium, Japan and Australia.
Pre-assignment Details: One subject was randomized to EVARREST, but instead received TachoSil; and analyzed in EVARREST ITT set and in TachoSil group for Safety set. Therefore, Safety set consists of 75 subjects in EVARREST arm and 81 subjects in TachoSil arm, while the ITT set consists of 76 subjects in EVARREST arm and 80 subjects in TachoSil arm.
Groups:
- EVARREST Fibrin Sealant Patch: EVARREST® Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin.
- TachoSil: TachoSil is a topical fibrin sealant patch consisting of human fibrinogen and human thrombin coated onto an equine collagen sponge.
Period: Overall Study
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Started | 75 | 81
Intent to Treat (Randomized Subjects) | 76 | 80
Completed | 70 | 77
Not Completed | 5 | 4
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data was summarized for the Safety Analysis Set, which consists of all subjects on whom the procedure was started.
Groups:
- Total: Total of all reporting groups
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil | Total
Number analyzed (Participants) | 75 | 81 | 156
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 < 50 years | 14 | 12 | 26
  50 < 65 years | 21 | 32 | 53
  65 < 75 | 22 | 25 | 47
  >= 75 | 18 | 12 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 56 | 61 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 68 | 76 | 144
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 62 | 66 | 128
  Black or African American | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Asian | 10 | 11 | 21
  Other | 1 | 1 | 2
BMI Category [Number; unit: Participants]
  Underweight | 2 | 0 | 2
  Normal | 20 | 18 | 38
  Overweight | 31 | 32 | 63
  Obese | 20 | 30 | 50
  Morbidly obese | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemostasis at the Target Bleeding Site (TBS) at 3 Minutes Following Treatment Application.
Description: Number of subjects achieving hemostasis at the Target Bleeding Site (TBS) at 3 minutes following treatment application, with no re-bleeding at the TBS any time prior to the initiation of final chest wall closure
Time Frame: Intraoperative, 3 minutes following treatment application
Population: The primary endpoint analysis was based on the Intent to Treat (ITT) analysis set, consisting of all randomized subjects.
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Number analyzed (Participants) | 76 | 80
Participants | 57 | 36
Statistical Analysis 1: Comparison: EVARREST Fibrin Sealant Patch vs TachoSil; Superiority; Test type: Superiority or Other; p = 0.0001, Adaptive group sequential design; Whitehead method for triangular test

2. Secondary Outcome: Number of Participants With Hemostasis at the Target Bleeding Site (TBS) at 6 Minutes Following Treatment Application
Description: The number of subjects achieving hemostatic success at 6 minutes following treatment application with no re-bleeding at the TBS any time prior to the initiation of final chest wall closure.
Time Frame: Intraoperative, 6 minutes following treatment application
Population: The secondary endpoint analyses were based on the Intent to Treat (ITT) analysis set.
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Number analyzed (Participants) | 76 | 80
Participants | 59 | 45
Statistical Analysis 1: Comparison: EVARREST Fibrin Sealant Patch vs TachoSil; Test type: Superiority or Other; p = 0.0046, Chi-squared

3. Secondary Outcome: Number of Participants With Hemostasis at the Target Bleeding Site (TBS) at 10 Minutes Following Treatment Application
Description: The number of subjects achieving hemostatic success at 10 minutes following treatment application, with no re-bleeding at the TBS any time prior to the initiation of final chest wall closure.
Time Frame: Intraoperative, 10 minutes following treatment application
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Number analyzed (Participants) | 76 | 80
Participants | 64 | 56

4. Secondary Outcome: Number of Participants With Re-bleeding at the Target Bleeding Site (TBS) Requiring Additional Treatment
Description: The number of subjects who, after the initial establishment of TBS hemostasis at 3 minutes, had intra-operative re-bleeding requiring treatment at the TBS
Time Frame: Intra-operative, prior initiation of final chest wall closure.
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Number analyzed (Participants) | 76 | 80
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: From surgical procedure through the 60 day follow-up (+/-14 days)
Arm/Group | EVARREST Fibrin Sealant Patch | TachoSil
Serious Adverse Events (participants affected / at risk) | 31/75 | 34/81
Other Adverse Events (participants affected / at risk) | 73/75 | 80/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVARREST Fibrin Sealant Patch (N=75) | TachoSil (N=81)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 8
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 3 | 0
Myocardial depression (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 3
Right ventricular failure (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 4 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 4
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
International normalised ratio fluctuation (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=75) | TachoSil (N=81)
Anaemia (Blood and lymphatic system disorders) | 18 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 7
Atrial fibrillation (Cardiac disorders) | 34 | 29
Cardiac failure congestive (Cardiac disorders) | 4 | 1
Pericardial effusion (Cardiac disorders) | 1 | 8
Tachycardia (Cardiac disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 15 | 15
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 19 | 20
Vomiting (Gastrointestinal disorders) | 5 | 7/75
Chest pain (General disorders) | 5 | 3
Oedema peripheral (General disorders) | 5 | 13
Pain (General disorders) | 9 | 11
Pyrexia (General disorders) | 11 | 10
Pneumonia (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 9 | 5
Wound infection (Infections and infestations) | 4 | 4
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 4 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 | 5
Procedural pain (Injury, poisoning and procedural complications) | 9 | 5
Wound complication (Injury, poisoning and procedural complications) | 3 | 9
Fluid overload (Metabolism and nutrition disorders) | 12 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 3
Dizziness (Nervous system disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 2 | 5
Confusional state (Psychiatric disorders) | 3 | 6
Delirium (Psychiatric disorders) | 3 | 7
Renal failure acute (Renal and urinary disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 1 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 24 | 22
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hypertension (Vascular disorders) | 4 | 9
Hypotension (Vascular disorders) | 15 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days